CLINICAL TRIAL: NCT00785577
Title: A Phase 2 Study of the Effects of LY545694, an iGluR5 Antagonist, in the Treatment of Subjects With Painful Diabetic Neuropathy.
Brief Title: A Study for Treatment of Pain in Patients With Diabetic Neuropathy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11977; H8C-MC-LQBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-04

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin; dasolampanel etibutil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): LY545694 placebo twice daily (BID) oral (po) for 5 weeks and pregabalin placebo capsules thrice daily (TID) po for 6 weeks
  Interventions: Drug: Placebo
- Pregabalin (Active Comparator): Pregabalin thrice daily (TID) oral for 6 weeks: 50 mg TID po for Week 1, 100 mg TID po for Weeks 2 - 5, and 50 mg TID po taper for Week 6
  LY545694 placebo BID po for 5 weeks
  Interventions: Drug: Pregabalin
- LY545694 21 mg (Experimental): LY545694 21 milligrams (mg) BID po for 1 week
  Pregabalin placebo TID po for 6 weeks
  Interventions: Drug: LY545694 21 mg
- LY545694 49 mg (Experimental): LY545694 escalated to 49 mg BID po during Week 2; possible titration down to 21 mg BID po within 1 week of escalation for remainder of study treatment.
  Pregabalin placebo TID po for 6 weeks
  Interventions: Drug: LY545694 49 mg
- LY545694 105 mg (Experimental): LY545694 escalated to 105 mg BID po during Week 3 through Week 5; possible titration down to 49 mg BID po within 1 week of escalation for the remainder of study treatment.
  Pregabalin placebo TID po for 6 weeks
  Interventions: Drug: LY545694 105 mg

INTERVENTIONS:
Drug: Placebo — LY545694 placebo BID po for 5 weeks
  Pregabalin placebo capsules TID po for 6 weeks
  Arms: Placebo
Drug: Pregabalin — Pregabalin TID po for 6 weeks: 50 mg TID po for Week 1, 100 mg TID po for Weeks 2 - 5, and 50 mg TID po taper for Week 6
  LY545694 placebo BID po for 5 weeks
  Arms: Pregabalin
Drug: LY545694 21 mg — LY545694 21 mg BID po for 1 week
  Pregabalin placebo TID po for 6 weeks
  Other Names: LY545694
  Arms: LY545694 21 mg
Drug: LY545694 49 mg — LY545694 escalated to 49 mg BID po for 1 week during Week 2.
  Pregabalin placebo TID po for 6 weeks.
  Other Names: LY545694
  Arms: LY545694 49 mg
Drug: LY545694 105 mg — LY545694 105 mg BID po for 5 weeks
  Pregabalin placebo TID po for 6 weeks
  Other Names: LY545694
  Arms: LY545694 105 mg

SUMMARY:
The purpose of this study is to test whether a new treatment will be safe and effective in treating pain. Patients with diabetic peripheral neuropathy will be included.

ELIGIBILITY:
Inclusion Criteria:

* Have pain due to peripheral neuropathy based on disease diagnostic criteria: must have Type 1 or Type 2 diabetes mellitus, pain must being in the feet, with relatively symmetrical onset, daily pain must be present for at least 6 months, and diagnosis must be confirmed by a score of at least 3 on Part B of the Michigan Neuropathy Screening Instrument.
* Have stable glycemic control, and glycated hemoglobin (HbA1c) less than or equal to 10%
* Mean score of at least 4 on the 24-hour average page severity assessment from (from daily diary) Visits 2 to 3.
* Fully completed daily diaries for at least 70% of the days between Visit 2 and 3.
* Women must test negative for a serum pregnancy test at Visit 1, and must agree to use medically acceptable and reliable means of birth control as determined by the investigator during the study and for 1 month following the last dose of study drug.
* Are competent and able to freely give own informed consent.
* Have an educational level and degree of understanding such that they can communicate intelligible with the investigator and study coordinator.
* Have been judged to be reliable and agree to keep all appointments for clinic visits, tests, and procedures required by the protocol.

Exclusion Criteria:

* Have historical exposure to drugs known to cause neuropathy, or a history of a medical condition, including pernicious anemia and hypothyroidism, that could have been responsible for neuropathy.
* Have pain that cannot be clearly differentiated from or conditions that interfere with the assessment of diabetic neuropathy pain.
* Have had treatment with any centrally active neuroleptic drug within 30 days of visit 3.
* Have had intolerance to pregabalin or have frequent and/or severe allergic reactions with multiple medications.
* Have current or previous (within the past 1 year) Axis 1 diagnosis of major depressive disorder, mania, bipolar disorder, psychosis, dysthymia, generalized anxiety disorder, alcohol or eating disorders according to Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria, as determined by the investigator and confirmed by the Mini-International Neuropsychiatric Interview (MINI).
* Have a serious of unstable cardiovascular, hepatic, renal, respiratory, ophthalmologic, gastrointestinal, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition that in the opinion of the investigator would compromise participation or be likely to lead to hospitalization during the course of the study.
* Have alanine aminotransaminase > 2 times upper limit of normal at Visit 1, based on reference ranges of central lab.
* Have prior renal transplant, current renal dialysis, or serum creatinine laboratory values > 1.5 times upper limit of normal, based on reference ranges of the central lab at Visit 1.
* Have a diagnosis or history of glaucoma.
* Are taking excluded medication that cannot be stopped and washed out prior to Visit 2.
* Have history of substance abuse or dependence within the past year, excluding nicotine and caffeine.
* Are judged clinically by the investigator to be at suicidal risk in the opinion of the investigator based upon clinical interview and the Columbia Suicide-Severity Rating Scale.
* Have a positive urine drug screen for any substance of abuse or excluded medication.
* Are unwilling or unable to comply with the use of a data collection device to directly record data from the subject (daily diary).
* Are pregnant or breast-feeding.
* Are investigator site personnel directly affiliated with this study and/or their immediate families.
* Are Lilly employees.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have a history of recurrent seizures other than febrile seizures.
* Have a history of severe gastroparesis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period 1 was an up to 5-week screening phase when participants stopped use of excluded medications (525 participants entered; 252 discontinued ). Study Period 2 was a 5-week, double-blind therapy period when randomization and dispensing of study drug occurred. Study Period 3 was a 1-week washout phase when all study medication was stopped.
Groups:
- Placebo: LY545694 placebo twice daily (BID) oral (po) for 5 weeks and pregabalin placebo capsules three times daily (TID) po for 6 weeks.
- Pregabalin: Pregabalin thrice daily TID po for 6 weeks: 50 mg TID po for Week 1, 100 mg TID po for Weeks 2 - 5, and 50 mg TID po taper for Week 6.
- LY545694 21 mg: LY545694 21 milligrams (mg) BID po for 1 week.
- LY545694 49 mg: LY545694 escalated to 49 mg BID po during Week 2; possible titration down to 21 mg BID po within 1 week of escalation for remainder of study treatment.
- LY545694 105 mg: LY545694 escalated to 105 mg BID po during Week 3 through Week 5; possible titration down to 49 mg BID po within 1 week of escalation for the remainder of study treatment.
Period: Study Period 2: Therapy Phase
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Started | 89 | 45 | 43 | 49 | 47
Completed | 78 | 36 | 25 | 36 | 27
Not Completed | 11 | 9 | 18 | 13 | 20
Not completed — Adverse Event | 5 | 7 | 14 | 10 | 17
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 1
Not completed — Entry Criteria Exclusion | 1 | 0 | 1 | 1 | 0
Not completed — Sponsor Decision | 1 | 0 | 1 | 1 | 0
Period: Study Period 3: 1-Week Washout Phase
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Started | 78 | 36 | 25 | 36 | 27
Completed | 78 | 36 | 25 | 35 | 26
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg | Total
Number analyzed (Participants) | 89 | 45 | 43 | 49 | 47 | 273
Age Continuous [Mean (Standard Deviation); unit: years] | 55.32 (10.00) | 56.89 (8.19) | 56.95 (8.35) | 58.59 (7.71) | 56.47 (7.77) | 56.62 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 17 | 20 | 25 | 19 | 118
  Male | 52 | 28 | 23 | 24 | 28 | 155
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 7 | 4 | 2 | 4 | 2 | 19
  Asian | 0 | 0 | 1 | 0 | 1 | 2
  Black or African American | 10 | 6 | 9 | 4 | 8 | 37
  Multiple | 1 | 0 | 1 | 1 | 1 | 4
  White | 71 | 35 | 30 | 40 | 35 | 211
Region of Enrollment [Number; unit: participants]
  United States | 57 | 29 | 28 | 29 | 28 | 171
  Mexico | 26 | 13 | 12 | 16 | 16 | 83
  Puerto Rico | 6 | 3 | 3 | 4 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Mean 24-hour Average Pain Severity (APS) Score at 5 Weeks
Description: This scale measured 24-hour APS scores. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). Least Squares (LS) Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: The analysis population was a modified intent-to-treat (ITT) population defined as participants who received either study drug with both baseline and at least 1 postbaseline measure. Last observation carried forward (LOCF) was conducted on the primary efficacy measure modified ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- LY545694 21 mg: LY545694 21 milligrams (mg) twice daily (BID) oral (po) for 1 week.
- LY545694 49 mg: LY545694 escalated to 49 mg twice daily (BID) oral (po) during Week 2; possible titration down to 21 mg BID po within 1 week of escalation for remainder of study treatment.
- LY545694 105 mg: LY545694 escalated to 105 mg twice daily (BID) oral (po) during Week 3 through Week 5; possible titration down to 49 mg BID po within 1 week of escalation for the remainder of study treatment.
Arm/Group | Placebo | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 78 | 26 | 35 | 30
units on a scale | -2.08 (0.22) | -2.22 (0.36) | -2.45 (0.32) | -2.42 (0.33)

2. Secondary Outcome: Change From Baseline in Weekly Mean Night Pain Severity Score at 5 Weeks
Description: This scale measured night pain APS scores. Data were recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: The analysis population was a modified intent-to-treat (ITT) population defined as participants who received either study drug with both baseline and at least 1 postbaseline measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 78 | 35 | 26 | 35 | 30
units on a scale | -2.31 (0.23) | -2.75 (0.33) | -2.25 (0.37) | -2.54 (0.33) | -2.21 (0.34)

3. Secondary Outcome: Change From Baseline in Weekly Mean Worst Daily Pain Severity Score at 5 Weeks
Description: This scale measured worst pain APS scores. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 78 | 35 | 26 | 35 | 30
units on a scale | -2.27 (0.25) | -2.87 (0.35) | -2.57 (0.40) | -2.77 (0.35) | -2.67 (0.37)

4. Secondary Outcome: Number of Participants With 30% Reduction in Weekly Mean 24-hour Average Pain Severity (APS) Score
Description: This scale measured the number of participants with a 30% reduction in weekly mean 24-hour APS score from baseline to endpoint. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline through 5 weeks
Population: The analysis population was a modified intent-to-treat (ITT) population defined as participants who received either study drug with both baseline and at least 1 postbaseline measure. LOCF was conducted on the primary efficacy measure modified ITT population.
Measure: Number; unit: participants
Arm/Group | Placebo | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 42 | 48 | 47
participants | 38 | 18 | 21 | 21

5. Secondary Outcome: Change From Baseline in Average Brief Pain Inventory - Interference (BPI-I) Subscale Score at 5 Weeks
Description: Average BPI-I measured self-reported degree of pain interference on function. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items. LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 37 | 26 | 35 | 30
units on a scale | -2.73 (0.25) | -2.81 (0.34) | -2.31 (0.39) | -2.73 (0.34) | -2.30 (0.36)

6. Secondary Outcome: Change From Baseline in Brief Pain Inventory - Severity (BPI-S) Subscale Score at 5 Weeks
Description: BPI-S measured self-reported severity of pain. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and current pain. LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 37 | 26 | 35 | 30
units on a scale
  BPI-S Worst Pain | -2.57 (0.29) | -3.54 (0.40) | -3.49 (0.47) | -2.94 (0.41) | -3.13 (0.44)
  BPI-S Least Pain | -1.76 (0.26) | -2.44 (0.35) | -1.99 (0.40) | -2.09 (0.36) | -1.54 (0.38)
  BPI-S Average Pain | -2.08 (0.26) | -2.92 (0.36) | -2.79 (0.41) | -2.50 (0.36) | -2.25 (0.38)
  BPI-S Current Pain | -2.44 (0.28) | -3.06 (0.38) | -2.66 (0.44) | -2.98 (0.39) | -2.51 (0.41)

7. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at 5 Weeks
Description: CGI-S measured severity of illness at the time of assessment compared with start of treatment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 37 | 26 | 35 | 30
units on a scale | -1.07 (0.11) | -1.02 (0.15) | -1.28 (0.18) | -1.07 (0.15) | -1.03 (0.16)

8. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Score at 5 Weeks
Description: PGI-I measured the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranged from 1 (very much better) to 7 (very much worse). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Week 5
Population: The analysis population was a modified intent to treat (ITT) population defined as participants who received either study drug with only postbaseline data collected.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 37 | 26 | 35 | 30
units on a scale | 2.58 (0.13) | 2.28 (0.18) | 2.37 (0.20) | 2.63 (0.18) | 2.41 (0.19)

9. Secondary Outcome: Change From Baseline in Short-form McGill Pain Questionnaire (SF-MPQ) Sensory Subscale Score at 5 Weeks
Description: SF-MPQ consisted of 11 sensory descriptors describing pain that were rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores were derived from the sum of the intensity rank values of the words chosen for sensory descriptors. The SF-MPQ sensory subscale was the sum of the 11 scores (ranged from 0 to 33, with 33 being the worst). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 36 | 26 | 35 | 30
units on a scale | -8.20 (0.73) | -8.60 (1.01) | -8.93 (1.20) | -8.95 (1.02) | -7.89 (1.10)

10. Secondary Outcome: Change From Baseline in Assessment of Sleep Questionnaire (ASQ) Total Score at 5 Weeks
Description: ASQ consisted of 21 items (including a single item to assess overall sleep quality) and 3 subscales: Sleep Onset and Maintenance (items 1-3, 5-6, 9, 11); Sleep Experience (items 4, 7, 8, 10, 12); and Awakening Experience (items 13-20). Each item was scored on a 5-point Likert scale, ranging from 0 (no sleep at all) to 5 (a lot of sleep). Each subscale was calculated as the mean of the individual items comprising the subscale. A total ASQ score was calculated as the mean of the subscale scores; higher scores represent better sleep.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 78 | 35 | 26 | 32 | 30
units on a scale | 0.76 (0.08) | 0.88 (0.11) | 0.67 (0.13) | 0.51 (0.12) | 0.55 (0.12)

11. Secondary Outcome: Change From Baseline in Neuropathy-Specific Quality of Life (NeuroQoL) Questionnaire Score at 5 Weeks
Description: NeuroQoL had 29 items: 13 assessed specific somatic experiences (pain, lost/reduced feeling, and diffuse sensory-motor symptoms); 14 assessed specific functional, social, and emotional experiences (restrictions in daily living activities, disruptions in social relationships, and emotional distress); 2 items assessed QoL and overall satisfaction. Items reported on a 5-point scale (never/not at all to all of the time/very much). Higher mean scores=more severe symptoms/greater disruption in functioning. First 27 items also associate with 3-point bothersome/importance scale (1=none to 3=very).
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 45 | 40 | 45 | 44
units on a scale | -0.56 (0.11) | -0.49 (0.15) | -0.58 (0.16) | -0.59 (0.15) | -0.31 (0.15)

12. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Health Survey Bodily Pain Score at 5 Weeks
Description: The SF-36 Health Status Survey was a generic, health-related scale assessing participants' quality of life on 8 domains (physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health) and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). MCS and PCS scores=0-100 (higher scores indicate better health status). Domain scores: general health=5-25; physical functioning=10-30; role-physical=4-8; role-emotional=3-6; social functioning=2-10; bodily pain=2-11; vitality=4-24; mental health=5-30.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 88 | 45 | 40 | 45 | 44
units on a scale | 7.51 (0.94) | 10.70 (1.26) | 8.16 (1.32) | 5.78 (1.24) | 6.33 (1.26)

13. Secondary Outcome: Change From Baseline of European Quality of Life Scale - 5 Dimensions (EQ-5D) at 5 Weeks: United States Population Based Index Score
Description: The EQ-5D was a generic, multidimensional, health-related, quality-of-life instrument. The profile allowed participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 was generated for each domain. For each participant, the outcome rating on the 5 domains was mapped to a single index through an algorithm. The index ranged between 0 and 1, with the higher score indicating a better health state perceived by the participant.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 88 | 45 | 40 | 45 | 44
units on a scale | 0.09 (0.02) | 0.09 (0.02) | 0.11 (0.02) | 0.05 (0.02) | 0.07 (0.02)

14. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Global Impairment Score at 5 Weeks
Description: The SDS was completed by the participant and was used to assess the effect of the participant's symptoms on work/social/family life. Total scores ranged from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 88 | 45 | 40 | 44 | 44
units on a scale | -2.96 (0.70) | -2.58 (0.94) | -2.63 (0.99) | -1.97 (0.95) | -3.04 (0.95)

15. Secondary Outcome: Number of Participants Who Discontinued Due to Adverse Events (AEs) During the Therapy (Double-blind) Phase and 1-Week Washout (Follow-up) Phase
Description: Participant discontinuation in the study due to serious and other non-serious AEs was measured during both the therapy (double-blind) phase and 1-week washout (follow-up) phase. A listing of serious and other non-serious AEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 6 weeks
Population: The safety analysis population included all 273 participants randomized to study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 45 | 43 | 49 | 47
participants
  Therapy (Double-blind) Phase | 5 | 7 | 14 | 10 | 17
  1-Week Washout (Follow-up) Phase | 0 | 0 | 0 | 1 | 1

16. Secondary Outcome: Number of Participants With Serious Treatment Emergent Abnormal High or Low Laboratory Values
Description: The number of participants by treatment group who had abnormal high or low laboratory values was reported by the investigator and summarized as serious adverse events (SAEs) from the "Investigations" system organ class during the treatment phase of the study. A listing of SAEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 5 weeks
Population: The safety analysis population included all 273 participants randomized to study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 45 | 43 | 49 | 47
participants
  Alanine aminotransferase (ALT) abnormal | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase (AST) abnormal | 0 | 0 | 0 | 0 | 1

17. Secondary Outcome: Change From Baseline in Vital Signs: Systolic Blood Pressure and Diastolic Blood Pressure at 5 Weeks
Description: Participants' systolic blood pressure and diastolic blood pressure were measured in millimeters of mercury (mmHg). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 37 | 26 | 35 | 30
millimeters of mercury (mmHg)
  Systolic Blood Pressure (mmHg) | -1.82 (1.37) | -3.18 (1.93) | 0.22 (2.26) | -0.24 (1.96) | 0.08 (2.10)
  Diastolic Blood Pressure (mmHg) | -0.87 (0.88) | -3.60 (1.25) | -0.07 (1.46) | 1.88 (1.26) | 0.77 (1.36)

18. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate at 5 Weeks
Description: Pulse rate was measured in beats per minute (bpm). LS Means were adjusted for baseline, investigator, treatment, visit, a treatment-by-visit interaction, and a baseline-by-visit interaction.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 37 | 26 | 35 | 30
beats per minute (bpm) | -1.06 (1.05) | -3.60 (1.49) | 0.87 (1.72) | 1.47 (1.51) | 1.66 (1.61)

19. Secondary Outcome: Number of Participants With Electrocardiogram Change in Heart Rate Using Bazett's (QTcB) and Fridericia's (QTcF) Formulas
Description: The number of participants having QTcF and QTcB change ≥ 30 msec was summarized.
Time Frame: Baseline through 5 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 78 | 41 | 36 | 42 | 36
participants
  QTcB ≥30 msec | 4 | 0 | 2 | 1 | 1
  QTcF ≥30 msec | 3 | 0 | 1 | 0 | 1

20. Secondary Outcome: Percentage of Participants With Reported Hypoglycemic Events
Description: Percentage of participants who reported hypoglycemic (lower than normal level of blood glucose) episodes was summarized as other non-serious adverse events (AEs) from the "Investigations" system organ class (preferred term = hypoglycemia). A listing of AEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 5 weeks
Population: The safety analysis population included all 273 participants randomized to study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 43 | 49 | 47
percentage of participants | 1.12 | 0.00 | 0.00 | 2.13

21. Secondary Outcome: Change From Baseline in Overall Total Quick Inventory of Depressive Symptomatology (QIDS) Score
Description: The QIDS was a 16-item patient-rated measure of depressive symptomatology. Each item had a 0 to 3 point scale. The total score ranged from 0 to 27 with higher scores indicative of greater severity. QIDS was calculated by summing the scores from the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) major depressive disorder criteria: depressed mood, loss of interest or pleasure, concentration/decision making, self outlook, suicidal ideation, energy/fatigability, sleep, weight/appetite change, and psychomotor changes.
Time Frame: Baseline, 5 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 45 | 43 | 49 | 47
units on a scale | -1.96 (0.22) | -1.49 (0.31) | -0.69 (0.34) | -0.46 (0.31) | 0.20 (0.32)

22. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal behaviors and ideations were provided. Suicidal behavior = a "yes" answer to any 1 of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation = a "yes" answer to any 1 of 5 suicidal ideation questions, which included the wish to be dead and 4 different categories of active suicidal ideation.
Time Frame: Baseline through week 5
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 45 | 43 | 49 | 47
participants
  Suicidal behaviors | 0 | 0 | 0 | 0 | 0
  Suicidal ideations | 1 | 0 | 1 | 0 | 1

23. Secondary Outcome: Number of Participants Reporting Blurry or Hazy Vision Using the Subjective Vision Inventory (SVI) Question 1 (Q1) at 5 Weeks
Description: This scale first asked if the participant was experiencing hazy or blurry vision or if he/she had difficulty focusing. If the answer was yes, follow-up questions rated the degree to which the issue impaired his/her ability to do work or to read.
Time Frame: Week 5
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 79 | 37 | 26 | 35 | 30
participants
  YES | 8 | 8 | 3 | 3 | 4
  NO | 71 | 29 | 23 | 32 | 26

24. Secondary Outcome: Pharmacokinetic (PK) Parameter: Clearance of LY545694 (CLp) and Compound 645838 (CLm)
Description: Clearance is the volume of plasma cleared of study drug LY545694 (CLp) and metabolite compound 645838 (CLm) per unit time. The original PK/pharmacodynamic (PD) relationship outcome measure analysis was not conducted; therefore, only PK data were reported.
Time Frame: Baseline through 5 weeks
Population: The PK dataset for population modeling consisted of quantifiable plasma LY545694 and Compound 64538 concentrations from participants following daily oral doses of LY545694 21 mg to LY545694 105 mg.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour (L/hr)
Groups:
- LY545694 Clearance (CLp): Plasma LY545694 concentrations were obtained following daily oral doses of LY545694 21 mg to LY545694 105 mg.
- Compound 645838 (CLm): Plasma Compound 645838 concentrations were obtained following daily oral doses of LY545694 21 mg to 105 mg.
Arm/Group | LY545694 Clearance (CLp) | Compound 645838 (CLm)
Number analyzed (Participants) | 115 | 118
Liters per hour (L/hr) | 79.1 [68.7 to 91.9] | 39.8 [35.8 to 44.8]

25. Secondary Outcome: Time to Response
Description: Time to response=first visit achieving a 30% reduction of weekly mean 24-hour APS score. Data were recorded daily (preferably at bedtime) on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). The number of days at which 50% of the participants at risk had at least 30% response was reported.
Time Frame: Baseline through 5 weeks
Population: as for outcome 2
Measure: Number; unit: time (days)
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 45 | 42 | 48 | 47
time (days) | 36 | 30 | 30 | 30 | 30

26. Secondary Outcome: Number of Participants With Neurological Treatment Emergent Adverse Events (TEAEs)
Description: The total number of TEAEs (serious and non-serious) that first occurred or worsened during the treatment period) from the "Nervous system disorders" system organ class was summarized. A listing of serious AEs (SAEs) and other non-serious AEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 5 weeks
Population: The safety analysis population included all 273 participants randomized to study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg
Number analyzed (Participants) | 89 | 45 | 43 | 49 | 47
participants | 17 | 22 | 16 | 24 | 23

ADVERSE EVENTS:
Groups:
- Pregabalin: Pregabalin thrice daily (TID) oral (po) for 6 weeks: 50 mg TID po for Week 1, 100 mg TID po for Weeks 2 - 5, and 50 mg TID po taper for Week 6
- Placebo Washout: A one-week washout period in which no placebo was taken.
- LY545694 21 mg Washout: A one-week washout period in which no LY545694 21 mg was taken.
- LY545694 49 mg Washout: A one-week washout period in which no LY545694 49 mg was taken.
- LY545694 105 mg Washout: A one-week washout period in which no LY545694 105 mg was taken.
- Pregabalin Washout: A one-week washout period in which no pregabalin was taken.
Arm/Group | Placebo | LY545694 21 mg | LY545694 49 mg | LY545694 105 mg | Pregabalin | Placebo Washout | LY545694 21 mg Washout | LY545694 49 mg Washout | LY545694 105 mg Washout | Pregabalin Washout
Serious Adverse Events (participants affected / at risk) | 0/89 | 1/43 | 1/49 | 1/47 | 0/45 | 0/89 | 0/43 | 0/49 | 1/47 | 0/45
Other Adverse Events (participants affected / at risk) | 53/89 | 33/43 | 43/49 | 40/47 | 31/45 | 15/89 | 4/43 | 7/49 | 7/47 | 6/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | LY545694 21 mg (N=43) | LY545694 49 mg (N=49) | LY545694 105 mg (N=47) | Pregabalin (N=45) | Placebo Washout (N=89) | LY545694 21 mg Washout (N=43) | LY545694 49 mg Washout (N=49) | LY545694 105 mg Washout (N=47) | Pregabalin Washout (N=45)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | LY545694 21 mg (N=43) | LY545694 49 mg (N=49) | LY545694 105 mg (N=47) | Pregabalin (N=45) | Placebo Washout (N=89) | LY545694 21 mg Washout (N=43) | LY545694 49 mg Washout (N=49) | LY545694 105 mg Washout (N=47) | Pregabalin Washout (N=45)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phosphenes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal exudates (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 3 (3) | 4 (4) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (12) | 12 (14) | 15 (17) | 12 (14) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (7) | 12 (13) | 8 (11) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram poor r-wave progression (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qrs complex prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grip strength decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monofilament pressure perception test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological examination abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Qrs axis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid factor increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salt craving (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased vibratory sense (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 8 (8) | 5 (8) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (13) | 1 (2) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyporeflexia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Narcolepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 3 (3) | 9 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 10 (11) | 7 (9) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 7 (7) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder sphincter atony (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Debridement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal stone removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin graft (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days